CLINICAL TRIAL: NCT00376168
Title: A Phase III, Multicenter, Randomized, Double-Blind Trial to Assess the Safety and Efficacy of Two Parallel Dose Groups of Plant Cell Expressed Recombinant Human Glucocerebrosidase (prGCD) in Patients With Gaucher Disease
Brief Title: A Phase III Trial to Assess the Safety and Efficacy of Plant Cell Expressed GCD in Patients With Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PB-06-001
Record Dates: First submitted 2006-09-12; First posted 2006-09-14 (Estimated); Results first posted 2012-07-26 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-09

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — taliglucerase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prGCD 30 Units/kg (Experimental)
  Interventions: Drug: Plant cell expressed recombinant glucocerebrosidase (prGCD)
- prGCD 60 Units/kg (Experimental)
  Interventions: Drug: Plant cell expressed recombinant glucocerebrosidase (prGCD)

INTERVENTIONS:
Drug: Plant cell expressed recombinant glucocerebrosidase (prGCD) — Intravenous infusion every two weeks for 9 months
  Other Names: Taliglucerase alfa
  Arms: prGCD 30 Units/kg
Drug: Plant cell expressed recombinant glucocerebrosidase (prGCD) — Intravenous infusion every 2 weeks for 9 months
  Other Names: Taliglucerase alfa
  Arms: prGCD 60 Units/kg

SUMMARY:
Gaucher disease, the most prevalent lysosomal storage disorder, is caused by mutations in the human glucocerebrosidase gene (GCD) leading to reduced activity of the lysosomal enzyme glucocerebrosidase and thereby to the accumulation of substrate glucocerebroside (GlcCer) in the cells of the monocyte-macrophage system.

This is the second trial to utilize a recombinant active form of lysosomal enzyme, glucocerebrosidase, (human prGCD) which is expressed and purified in a bioreactor system from transformed carrot plant root cell line.

DETAILED DESCRIPTION:
This will be a multi-center, randomized, double-blind, parallel group, dose-ranging trial to assess the safety and efficacy of prGCD in 30 untreated patients with Gaucher disease. Patients will receive IV infusion of prGCD every two weeks at the selected medical center. The duration of the study will be nine months. At the end of the 9-month treatment period (20 visits, 38 weeks) eligible patients will be offered enrollment in an open-label extension study.

There will be two treatment groups, 15 patients in each treatment group.

Treatment Group I: 30 units/kg every 2 weeks. Treatment Group II: 60 units/kg every 2 weeks.

All patients will have pharmacokinetic data collected over approximately 3 hours with frequent blood samples following the first and final doses of prGCD.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years or older
* Confirmed enzymatic diagnosis of Gaucher disease
* Splenomegaly defined as greater than eight times the expected volume (measured volume divided by estimated volume (0.2% of body weight)] as determined by MRI volumetric analysis
* Female patients of child-bearing potential who agree to use a medically acceptable method of contraception
* Thrombocytopenia (defined as platelet counts below the lower limit of normal) and/or anemia (defined by hemoglobin level at least 1 g/dL below normal range according to sex and age).
* Patients who have not received ERT in the past or patients whoc have not received ERT in the past 12 months and have a negative anti-glucocerebrosidase antibody test.
* Patients who have not received substrate reduction therapy (SRT) in the past 12 months.
* Ability to provide a written informed consent.

Exclusion Criteria:

* Currently taking another experimental drug for any condition
* Pregnant or nursing
* Presence of HIV and/or, HBsAg and/or hepatitis C infections
* Presence of severe neurological signs and symptoms, defined as complete ocular paralysis, overt myoclonus or history of seizures, characteristic of neuronopathic Gaucher disease.
* Previous anaphylactoid reaction to Cerezyme® or Ceredase®.
* History of allergy to carrots.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2007-08; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - University Research Foundation for Lysosomal Storage Diseases, Coral Springs, Florida
  - Division of Medical Genetics, Emory University School of Medicine, Decatur, Georgia
  - New York University Medical Center, New York, New York
- Mount Sinai Hospital, Toronto, Ontario, Canada
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- Israel (2):
  - Rambam Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
- Universita "La Sapienza", Rome, Italy
- Morningside Medi-Clinic, Morningside, South Africa
- Hospital Universitario Miguel Servet, Zaragoza, Spain
- Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Derived] Abbas R, Park G, Damle B, Chertkoff R, Alon S. Pharmacokinetics of Novel Plant Cell-Expressed Taliglucerase Alfa in Adult and Pediatric Patients with Gaucher Disease. PLoS One. 2015 Jun 8;10(6):e0128986. doi: 10.1371/journal.pone.0128986. eCollection 2015. PMID 26053270
- [Derived] Zimran A, Brill-Almon E, Chertkoff R, Petakov M, Blanco-Favela F, Munoz ET, Solorio-Meza SE, Amato D, Duran G, Giona F, Heitner R, Rosenbaum H, Giraldo P, Mehta A, Park G, Phillips M, Elstein D, Altarescu G, Szleifer M, Hashmueli S, Aviezer D. Pivotal trial with plant cell-expressed recombinant glucocerebrosidase, taliglucerase alfa, a novel enzyme replacement therapy for Gaucher disease. Blood. 2011 Nov 24;118(22):5767-73. doi: 10.1182/blood-2011-07-366955. Epub 2011 Sep 6. PMID 21900191
- [Derived] Winckler T. [Enzyme replacement therapy for Gaucher's Disease]. Pharm Unserer Zeit. 2008;37(5):352-3. doi: 10.1002/pauz.200890067. No abstract available. German. PMID 18729283

RESULTS

PARTICIPANT FLOW:
Groups:
- ELELYSO 30 Units/kg: Taliglucerase alfa 30 Units/kg by intravenous infusion every two weeks
- ELELYSO 60 Units/kg: Taliglucerase alfa 60 Units/kg by intravenous infusion every two weeks
Period: Overall Study
Arm/Group | ELELYSO 30 Units/kg | ELELYSO 60 Units/kg
Started | 16 | 16 (One patient randomized but not treated)
Completed | 14 | 15
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Pregnancy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ELELYSO 30 Units/kg | ELELYSO 60 Units/kg | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 16 | 31
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (11.8) | 36.0 (12.2) | 36.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 8 | 8 | 16
Region of Enrollment [Number; unit: participants]
  Canada | 1 | 1 | 2
  Spain | 0 | 1 | 1
  Chile | 1 | 1 | 2
  South Africa | 1 | 1 | 2
  Israel | 6 | 6 | 12
  Italy | 1 | 1 | 2
  United Kingdom | 0 | 1 | 1
  Mexico | 4 | 2 | 6
  Serbia | 2 | 2 | 4
Spleen Volume [Mean (Standard Deviation); unit: mL] — Measured by MRI
  mL | 2130.94 (1154.72) | 2117.38 (1356.17) | 2120 (1200)
Liver Volume [Mean (Standard Deviation); unit: mL] — Measured by MRI
  mL | 2880.60 (736.12) | 2481.31 (452.74) | 2600 (600)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] — Measured in central laboratory
  g/dL | 12.2 (1.7) | 11.4 (2.6) | 12 (2)
Platelet Count [Mean (Standard Deviation); unit: count/mm^3] — Measured in local laboratory
  count/mm^3 | 75,320 (40,861) | 65,038 (28,668) | 70,000 (32,000)
Chitotriosidase [Mean (Standard Deviation); unit: nmol/ml/hr] — Gaucher disease biomarker
  nmol/ml/hr | 28158 (11686) | 24702 (17428) | 26000 (14000)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Spleen Volume Measured by MRI.
Description: Calculated as percent change in spleen volume from Baseline to 9 months
Time Frame: Baseline and 9 months
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | ELELYSO 30 Units/kg | ELELYSO 60 Units/kg
Number analyzed (Participants) | 15 | 16
percentage of change | -26.91 (7.79) | -38.01 (9.38)
Statistical Analysis 1: Comparison: ELELYSO 30 Units/kg; The primary efficacy analysis was based on two one-sample t-tests (one for each treatment group) to determine if the percent change in spleen volume is different than zero. With 12 patients in each treatment group, there was greater than 95% power to detect a change of 20% or more using a one-sample t-test (alpha=0.025, 2-sided test to allow for each group to be tested separately) to evaluate the primary outcome of percent change in spleen volume after nine months; Test type: Superiority or Other; p < 0.0001, one-sample t-test; one-sample t-test (combined) to test the null hypothesis that percent change = 0
Statistical Analysis 2: Comparison: ELELYSO 60 Units/kg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, one-sample t-test — threshold for statistical significance = 0.025; one-sample t-test (combined) to test the null hypothesis that percent change = 0

2. Secondary Outcome: Change From Baseline in Liver Volume
Description: Calculated as percent change in liver volume from Baseline to 9 months
Time Frame: Baseline and 9 months
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | ELELYSO 30 Units/kg | ELELYSO 60 Units/kg
Number analyzed (Participants) | 15 | 16
percentage of change from baseline | -10.48 (11.27) | -11.11 (6.68)
Statistical Analysis 1: Comparison: ELELYSO 30 Units/kg; For each of the secondary endpoints, a one-sample t-test (% change in liver volume, mean change in hemoglobin and platelet count) was examined first for each dose using the step-down approach. Next, a mixed effects model that included dose and time, with subject as a random effect, was fit to examine whether there was a difference between dose groups, for those outcomes that were tested in the step-down approach; Test type: Superiority or Other; p = 0.0041, One-sample t-test
Statistical Analysis 2: Comparison: ELELYSO 60 Units/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, One-sample t-test

3. Secondary Outcome: Change in Hemoglobin
Description: Absolute change in Hemoglobin concentration from Baseline to Month 9
Time Frame: Baseline and Month 9
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | ELELYSO 30 Units/kg | ELELYSO 60 Units/kg
Number analyzed (Participants) | 14 | 16
g/dL | 1.6 (1.4) | 2.2 (1.4)
Statistical Analysis 1: Comparison: ELELYSO 30 Units/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0010, One-sample t-test
Statistical Analysis 2: Comparison: ELELYSO 60 Units/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, One-sample t-test

4. Secondary Outcome: Change in Platelet Count
Description: Change in Platelet count from Baseline to Month 9
Time Frame: Baseline and Month 9
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: count/mm^3
Arm/Group | ELELYSO 30 Units/kg | ELELYSO 60 Units/kg
Number analyzed (Participants) | 15 | 16
count/mm^3 | 11,427 (20,214) | 41,494 (47,063)
Statistical Analysis 1: Comparison: ELELYSO 30 Units/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0460, One-sample t-test
Statistical Analysis 2: Comparison: ELELYSO 60 Units/kg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0031, One-sample t-test

5. Other Pre Specified Outcome: Change in Chitotriosidase
Description: Change in Chitotriosidase from Baseline to Month 9
Time Frame: Baseline and Month 9
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: nmol/ml/hr
Arm/Group | ELELYSO 30 Units/kg | ELELYSO 60 Units/kg
Number analyzed (Participants) | 14 | 15
nmol/ml/hr | -14,548 (8,025.8) | -12,538 (14,489)

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | ELELYSO 30 Units/kg | ELELYSO 60 Units/kg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 6/16 | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ELELYSO 30 Units/kg (N=16) | ELELYSO 60 Units/kg (N=16)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Glycosuria (Renal and urinary disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No